CLINICAL TRIAL: NCT07353840
Title: T Cell Lymphoma -Stratified Therapy After Response to First-line Treatment-CR
Acronym: T-START-CR
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SHSYXYK-PTCL-CR-prospective
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Peripheral T Cell Lymphoma; autologous hematopoietic stem cell transplantation; observation; complete response
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Pathologic Complete Response | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation: This is a patient cohort that receives monitoring after first-line therapy with complete response.
  Interventions: Other: Observation
- Auto-HSCT: Auto-HSCT involves the infusion of the patient's own previously collected stem cells.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Auto-HSCT involves the infusion of the patient's own previously collected stem cells.
  Groups: Auto-HSCT
Other: Observation — This is a patient cohort that receives monitoring after first-line therapy with complete response.
  Groups: observation

SUMMARY:
This study is a multicenter, two-arm, prospective clinical trial, comprising two groups: the observation group and the autologous hematopoietic stem cell transplantation group (Auto-HSCT). It aims to evaluate the efficacy and safety of Auto-HSCT and observation in the treatment of peripheral T-cell lymphoma that has achieved complete response (CR) after first-line therapy. During the screening/baseline period, informed consent will be obtained, and inclusion/exclusion criteria will be verified. Group assignment (Observation vs. Auto-HSCT) will be determined taking into account the patient's preference. The study plans to enroll 80 patients in each group. Data on demographics and medical history will be collected, and assessments including vital signs, physical examination, PET-CT, bone marrow aspiration smear, flow cytometry, and bone marrow pathology will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years (inclusive) at the time of signing the Informed Consent Form (ICF).
2. ECOG Performance Status score of 0 or 1, with no deterioration over the preceding two weeks.
3. Life expectancy of at least 12 weeks.
4. Histologically confirmed diagnosis of PTCL by the central study site according to the 2016 revised WHO classification of lymphoid neoplasms (Swerdlow SH et al. 2016). Eligible histological subtypes are restricted to the following:

   1. Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS)
   2. Anaplastic large cell lymphoma, ALK-negative (ALK- ALCL)
   3. Follicular helper T-cell lymphoma or PTCL with a TFH phenotype (FTCL or PTCL-TFH)
5. Must have achieved a Complete Response (CR) as assessed per the Lugano 2014 classification criteria for lymphoma response after first-line systemic standard therapy (CHOP or a CHOP-like regimen).
6. Adequate hepatic and renal function, defined as:

   1. Hepatic: Serum total bilirubin ≤ 2 × ULN (or ≤ 3.0 × ULN in cases of Gilbert's syndrome or documented baseline liver involvement); Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 × ULN (or ≤ 5.0 × ULN in cases of liver involvement).
   2. Renal: Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min as calculated by the Cockcroft-Gault formula or measured.
7. Left Ventricular Ejection Fraction (LVEF) ≥ 50% as measured by Multigated Acquisition (MUGA) scan or Echocardiography (ECHO).
8. Voluntary participation in the clinical study; full understanding and awareness of the study, and having signed the ICF; willingness and ability to comply with and complete all trial procedures.

Exclusion Criteria:

1.Ann Arbor Stage I disease. 2.History of any other malignancy within the past 5 years, except for locally curable malignancies that have been treated with curative intent (e.g., basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast).

3.Active infection, including:

1. Known active or latent tuberculosis, evidenced by a positive tuberculin (PPD) skin test (where a positive result is defined as an induration >10 mm or per local clinical standards) or findings suggestive of active/latent TB on chest X-ray/CT.
2. Known history of Human Immunodeficiency Virus (HIV) infection and/or AIDS.
3. Chronic active hepatitis B or C infection:

   1. For hepatitis B virus (HBV): Subjects who are HBV DNA positive are excluded. Subjects with undetectable HBV DNA levels are eligible. The upper limit of normal (ULN) for HBV DNA is determined by the local laboratory at each center.
   2. For hepatitis C virus (HCV): Subjects who are HCV RNA positive are excluded. Subjects with undetectable HCV RNA are eligible. The ULN for HCV RNA is determined by the local laboratory at each center.
4. Active viral infections other than hepatitis B or C (e.g., herpes zoster), or cytomegalovirus (CMV) infection.
5. Infection requiring intravenous antimicrobial therapy: evidenced by infection-related hemodynamic instability, worsening or new-onset infectious symptoms/signs, radiologic evidence of a new infectious focus, or persistent fever without localizing signs where infection cannot be ruled out.
6. Positive serological test for Epstein-Barr virus (EBV). 4.Poorly controlled cardiac symptoms or diseases, such as: i. Heart failure > New York Heart Association (NYHA) Class II. ii. Unstable angina. iii. Myocardial infarction within the past year. iv. Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.

5.Pregnant or lactating women, and subjects of childbearing potential unwilling to employ effective contraception.

6.Patients with psychiatric disorders or those unable to provide informed consent.

7.Any other condition which, in the investigator's judgment, makes the subject unsuitable for participation in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with peripheral T-cell lymphoma that has achieved complete response (CR) after first-line therapy.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
event-free survival (EFS) | up to 2 years for the 2y-EFS
  Event-free survival (EFS) rates post-transplant. An event is defined as whichever of the following occurs first: disease progression, death from any cause, commencement of new anti-tumor therapy, or a treatment-related serious adverse event (specifically including disabling events or secondary neoplasms). Subjects who were event-free at the data cutoff will be censored on the date of their last tumor assessment.

SECONDARY OUTCOMES:
1y and 2y-cumulative relapse rates (CIR) | up to 1 years for the 1y-CIR and up to 2 years for the 2y-CIR
  The cumulative probability of disease progression (including relapse or progression of the primary disease) within 1 or 2 years after transplantation, with non-progression-related death treated as a competing event.
Disease-Free Survival (DFS) | up to 1 years for the DFS
  DFS means the time from transplantation until the first occurrence of any of the following events: disease recurrence, disease progression, or death from any cause.
overall survival (OS) | up to 1 years for the 1y-OS and up to 2 years for the 2y-OS
  The probability of survival at 1 or 2 years, measured from the date of transplantation to death from any cause. Patients who are still alive at the time of analysis will be censored on the last follow-up date.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tournilhac O, Altmann B, Friedrichs B, Bouabdallah K, Leclerc M, Cartron G, Turlure P, Reimer P, Wagner-Drouet E, Sanhes L, Houot R, Roussel M, Kroschinsky F, Dreger P, Viardot A, de Leval L, Rosenwald A, Gaulard P, Wulf G, Villate A, Latiere C, Elmaagacli A, Glass B, Poeschel V, Damaj G, Sibon D, Durot E, Bilger K, Banos A, Haenel M, Dreyling M, Keller U, Tiab M, Drenou B, Cornillon J, Nguyen S, Robin M, Nickelsen M, Trumper L, Lenz G, Ziepert M, Schmitz N; French Lymphoma Study Association (LYSA), the Societe Francophone de greffe de moelle et Therapie Cellulaire (SFGM-TC), and the German Lymphoma Alliance (GLA). Long-Term Follow-Up of the Prospective Randomized AATT Study (Autologous or Allogeneic Transplantation in Patients With Peripheral T-Cell Lymphoma). J Clin Oncol. 2024 Nov 10;42(32):3788-3794. doi: 10.1200/JCO.24.00554. Epub 2024 Sep 13. PMID 39270145
- [Background] Schmitz N, Truemper L, Bouabdallah K, Ziepert M, Leclerc M, Cartron G, Jaccard A, Reimer P, Wagner E, Wilhelm M, Sanhes L, Lamy T, de Leval L, Rosenwald A, Roussel M, Kroschinsky F, Lindemann W, Dreger P, Viardot A, Milpied N, Gisselbrecht C, Wulf G, Gyan E, Gaulard P, Bay JO, Glass B, Poeschel V, Damaj G, Sibon D, Delmer A, Bilger K, Banos A, Haenel M, Dreyling M, Metzner B, Keller U, Braulke F, Friedrichs B, Nickelsen M, Altmann B, Tournilhac O. A randomized phase 3 trial of autologous vs allogeneic transplantation as part of first-line therapy in poor-risk peripheral T-NHL. Blood. 2021 May 13;137(19):2646-2656. doi: 10.1182/blood.2020008825. PMID 33512419